CLINICAL TRIAL: NCT00740337
Title: Specialized Center of Clinically Oriented Research: Alveolar and Airway Mechanisms of COPD. Airway Determinants: Innate Immune Signaling (Project 4)
Brief Title: Factors That Affect the Development of COPD Symptoms
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 582
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Natural Killer T-cell; Interleukin-13; Innate Immune Signaling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, isolated RNA and DNA, lung tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD: Participants in this group will be people who have COPD and plan to undergo lung resection surgery at Barnes-Jewish Hospital (BJH).
- Control: Participants in this group will be people who do not have COPD and plan to undergo lung resection surgery at BJH.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the fourth most common cause of death in the United States. There is no cure and the disease gets worse over time. Although it usually occurs in people who smoke cigarettes, researchers do not know exactly how smoking leads to COPD. This study will compare blood and tissue samples from smokers and nonsmokers with and without COPD to determine why some COPD symptoms occur in some people and not others.

DETAILED DESCRIPTION:
COPD is a chronic lung disease in which the lungs' airways and balloon-like air sacs, called alveoli, are damaged, lose their shape, and become floppy. As a result, they cannot fully inflate to allow the maximum amount of air through. COPD is usually the result of many years of cigarette smoking. Breathing in other kinds of lung irritants, such as pollution, dust, or chemicals, over a long period of time may also cause or contribute to COPD. Some people with COPD have an excess of mucus in their lungs, possibly caused by an overactive immune response, which can lead to coughing and shortness of breath. Although cigarette smoking seems to make this symptom worse, researchers are not sure why it occurs in some people and not others. This study will examine and compare blood and lung tissue samples from smokers and nonsmokers with and without COPD to determine what physiological differences, environmental factors, genes, and biomarkers contribute to the development of and symptoms associated with COPD.

Before their scheduled lung resection surgery, participants in this study will attend one study visit. It will last approximately 1 to 2 hours and will consist of answering questions about medical history, filling out health questionnaires, and providing a blood sample. After the surgery, study researchers will take the lung tissue that was removed and examine it in a laboratory. Participants will be contacted by study staff if, when examining the lung tissue, researchers discover that a participant has a medical disorder that current treatment can stop or improve. Also, participants will be contacted at the end of the study to answer brief questions about their health.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in English
* Able to participate in the informed consent process
* Planned lung resection at BJH
* Acceptable pulmonary function tests done at BJH within 1 month of enrollment
* Acceptable chest CT scan done at BJH within 3 years of enrollment

Exclusion Criteria:

* Pregnant
* Prisoner
* Vulnerable populations
* Clinically significant lung disease other than COPD and the indication for resection (e.g., cystic fibrosis, bronchiectasis, obliterative bronchiolitis, airway lesion)
* Coexisting active chronic inflammatory or collagen vascular disease, immune deficiency of any kind, or previous organ transplant
* Known active hepatitis B, hepatitis C, or HIV/AIDS (not prospectively evaluated)
* Systemic chemotherapy within past 1 month (30 days)
* Hematologic malignancy or thoracic radiation within past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People in this study will be invited to participate if they plan to undergo lung resection surgery at BJH.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Holtzman, MD, Principal Investigator — Pulmonary and Critical Care, Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States